CLINICAL TRIAL: NCT02754960
Title: A Randomised, Double-blind, Placebo-controlled Study of Thalidomide in Gastrointestinal Vascular Malformation Related Bleeding
Brief Title: Efficacy Study of Thalidomide in Gastrointestinal Vascular Malformation Related Bleeding
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhizheng Ge, the director of the endoscopy center, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rjyyxhk57809
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Gastrointestinal Hemorrhage; Vascular Malformation
Keywords: Gastrointestinal bleeding; Vascular malformation; Angiodysplasia; Thalidomide
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Vascular Malformations; Angiodysplasia | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide group (Active Comparator): Patients were randomly assigned to the thalidomide group and received 100 mg of thalidomide (Pharmaceutical Co., Ltd. of Chang Zhou, China) orally four times daily at 10 p.m. for four months.
  Interventions: Drug: Thalidomide
- Placebo group (Placebo Comparator): Patients were randomly assigned to the placebo group and received 100 mg of thalidomide placebo (Pharmaceutical Co., Ltd. of Chang Zhou, China) orally four times daily at 10 p.m. for four months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thalidomide — Interventions administered (dosage, 100mg; dosage form, 25mg; frequency of administration, 1 time daily at 10 p.m)
  Other Names: Softenon
  Arms: Thalidomide group
Drug: Placebo — Placebo administered (dosage, 100mg; dosage form, 25mg; frequency of administration, 1 time daily at 10 p.m)
  Other Names: Thalidomide placebo
  Arms: Placebo group

SUMMARY:
Background: Repeated bleeding from gastrointestinal vascular malformations remains to be a major therapeutic challenge.

Methods: The investigators performed a randomised, double-blind, placebo-controlled, single centre study to assess the long-term efficacy and safety of thalidomide 100mg qn p.o. or placebo 100 mg qn p.o. administration for 4 months in subjects with recurrent gastrointestinal bleeding due to vascular malformations. Patients with at least six episodes of bleeding in the prior year due to vascular malformation were randomly grouped, prescribed a four-month regimen of either 100mg of thalidomide or 100 mg of placebo orally one time daily, and monitored for at least one year. The primary end point was defined as the patients whose rebleeds decreased from baseline by ≥ 50% at 12 months. Rebleeding was defined based on a positive fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) at any visit after treatment. Secondary outcomes included the changes from baseline in participants dependent on blood transfusions and transfused packed red cell units, bleeding episodes, bleeding durations, and hemoglobin levels at 12 months. Statistical significance was defined at P < 0.05.

DETAILED DESCRIPTION:
Study design:

The study will be carried out as a single-centre, randomized, double-blind, parallel-group, placebo-controlled phase II study in subjects with recurrent gastrointestinal bleeding due to vascular malformations.

Subjects Enrollment and Assignment:

Approximately 100 patients aged between 40-85 years with recurrent gastrointestinal bleeding (melena and/or fresh hematemesis or positive FOBT) at least 6 times within one year, verified as vascular malformation by capsule endoscopies or enteroscopies at baseline.

Randomization was performed through the proc plan procedure of SAS, using the method of randomly permuted blocks of 4. Within each block, the number of patients allocated to each of the two treatments was equal. Subjects who are eligible for randomisation will be given a subject number in consecutive order within blocks, and the investigational products packed corresponding to this number. The subject will be allocated to one of the two treatment groups, i.e. Thalidomide and placebo, according to a computer generated list provided by Pharmaceutical Co., Ltd. of Chang Zhou, China. If a subject discontinues from the study, the subject number will not be reused, and the subject will not be allowed to re-enter the study.

Intervention:

The included patients were prospectively randomized into two groups: the thalidomide group and the placebo group (Thalidomide group: Thalidomide p.o. 100 mg for 4 months, qn; Placebo group: Placebo for thalidomide p.o. 100 mg for 4 months, qn).

The following concomitant medications are not allowed during the study as they interfere with the disease under study: Anti-angiogenic agents or other putative immunomodulators, Anti-platelet drugs, anticoagulants, or Chinese medications (with salicylates), gingko, or Echinacea, Somatostatin Heparin, Warfarin (including other Vit K antagonists), NSAIDs(including low dose); or as there is a potential risk for drug-drug interactions: Paxil (paroxetine), Mysoline (primidone), Keppra (levetiracetam), Plaquenil (hydroxychloroquine), St John's Wort (st. john's wort), Tegretol (carbamazepine), Zometa (zoledronic acid).

Assessment of response and adverse events:

The primary end point was defined as the patients whose rebleeds decreased from baseline by ≥ 50% at 12 months. Rebleeding was defined based on a positive fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) at any visit after treatment. The secondary outcomes included the changes from baseline in participants dependent on blood transfusions and transfused packed red cell units, bleeding episodes, bleeding durations, and hemoglobin levels at 12 months.

An adverse event (AE) is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.

A serious adverse event is an AE occurring during any study phase (ie, run-in, treatment, follow-up), and at any dose of the investigational product, comparator or placebo, that fulfils one or more of the following criteria:

Results in death; Deep vein thrombosis (DVT); Is immediately life-threatening; Requires prolongation of existing hospitalisation; Results in persistent or significant disability or incapacity; Is a congenital abnormality or birth defect; Is an important medical event that may jeopardise the subject or may require medical intervention to prevent one of the outcomes listed above.

Evaluation of Patients and Follow-up:

* Certified research nurses collected information on the demographics and medical and social histories of all patients enrolled in the study.
* After screening and baseline evaluations, the patients were closely monitored in the hospital for at least one week. They were then followed twice monthly during the four-mouth course of treatment and once a month thereafter.
* Clinical follow-up was performed by qualified doctors. At all visits, the bleeding-related parameters (number and duration), a physical examination was performed and laboratory values were obtained for FOBT, complete blood counts, serum chemistries, and hepatic and renal function. Neuropathy and other adverse events were also assessed.
* Patients were advised to refrain from any other non-prescribed medicines, especially rebleeding-related medications such as aspirin, NSAIDs, anti-platelet drugs, anticoagulants, and Chinese medications (with salicylates), gingko, or Echinacea.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-85 years; women were post-menopausal, post-tubal ligation, or on some form of birth control like long-term laying up contraceptive ring or using condom;
* History of at least six documented gastrointestinal bleeding episodes in the year prior to randomization, which were refractory or inaccessible to endoscopic therapy or surgical ectomy;
* Confirmed diagnosis of vascular malformation by esophagogastroduodenoscopy (EGD), capsule endoscope (CE), double-balloon endoscope (DBE), or colonoscopy, but no obvious infectious, neoplastic, or other specific diagnosis;
* Angiodysplasia at endoscopy characterized by focal or diffused venous/capillary lesions presenting as bright red ectatic vessels or pulsatile red protrusions, with surrounding venous dilatation or patchy erythema with or without oozing;

Exclusion Criteria:

* Less than 1 year of bleeding history;
* GI bleeding caused by Esophageal varices, Mallory Weiss syndrome, Zollinger-Ellison syndrome, Suspicion of gastric malignancy at baseline endoscopy, Post-Billroth-resection, Biliary disorders, Gastrointestinal tumors, Crohn's disease or Ulcerative colitis, Hemangioma or unknown source of GI bleeding;
* Bleeding that needs emergent endoscopic treatment or surgery;
* Any significant "alarm symptoms" within the past 6 months, such as, unintentional weight loss, signs of gastrointestinal bleeding more than 2 weeks prior to enrolment, jaundice, or any other sign indicating serious or malignant disease;
* Malignancy or clinically significant cardiovascular, pulmonary, renal, pancreatic, hepatic disease, cirrhotic or portal hypertension gastropathy, rheumatologic disorders, uncontrollable diabetes mellitus or hypertension as judged by the investigator;
* A history of severe bilateral peripheral neuropathy or seizure activity, thromboembolic disease;
* A history of treatment with any dose of systemic or oral topical corticosteroids or aspirin, NSAIDs, anti-platelet drugs, anticoagulants, or Chinese medications (with salicylates), gingko, or Echinacea, or other putative immunomodulators or anti-angiogenic agents;
* Haemorrhagic disorders, platelets<100 x 109/ L, APTT>1.5x upper limit of normal (ULN), or treatment with low-molecular weight heparin;
* Need for continuous concurrent therapy during the study period with NSAIDs, ASA (including low dose),Warfarin (including other Vit K antagonists), anti-platelet drugs, anticoagulants, mephenytoin, atazanavir or Chinese medications (with salicylates), gingko, or Echinacea, or other putative immunomodulators or anti-angiogenic agents;
* Pregnancy or lactation. Woman of child-bearing potential must be either non-pregnant or postmenopausal or must use a reliable form of contraception during the study period, as judged by the investigator;
* Allergy to study medications;
* Currently undergoing systemic cancer chemotherapy or receiving radiation or had underwent systemic cancer chemotherapy or received radiation treatment.
* Use of any other investigational compound or participation in another clinical trial within 30 days prior to start of study medication;
* Alcohol and/or drug abuse (addiction or drug dependence) or any condition associated with poor compliance, including expected non-cooperation, as judged by the investigator;
* Previous participation in the study;
* Involvement in the planning and conduct of the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects whose bleeding episode decreased from baseline by ≥ 50% at 12 months follow-up after 4-month treatment | 12 months
  Proportion of subjects whose bleeding episode decreased from baseline by ≥ 50% at 12 months follow-up after 4-month treatment. The details are showed as follows: Reduction of bleeding episode = [(total bleeding episodes at 12 months - total bleeding episodes at a year before randomisation)/total bleeding episodes at a year before randomisation (baseline)]*100%. Rebleeding was defined based on a positive fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) at any visit after treatment.

SECONDARY OUTCOMES:
Change from baseline in bleeding episodes at 12 months | baseline and 12 months
  Change from baseline in bleeding episodes at 12 months
Change from baseline in bleeding duration at 12 months | baseline and 12 months
  Change from baseline in bleeding duration at 12 months
Change from baseline in proportion of subjects who dependent on blood transfusions at 12 months | baseline and 12 months
  Change from baseline in proportion of subjects who dependent on blood transfusions at 12 months
Change from baseline in number of blood units transfused in subjects who dependent on blood transfusions at 12 months | baseline and 12 months
  Change from baseline in number of blood units transfused in subjects who dependent on blood transfusions at 12 months
Change from baseline in average hemoglobin (Hb) level at 12 months | baseline and 12 months
  Change from baseline in average hemoglobin (Hb) level at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhizheng Ge, Ph.D, MD., Principal Investigator — Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Gastroenterology department; Ren Ji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Jacobson JM, Greenspan JS, Spritzler J, Ketter N, Fahey JL, Jackson JB, Fox L, Chernoff M, Wu AW, MacPhail LA, Vasquez GJ, Wohl DA. Thalidomide for the treatment of oral aphthous ulcers in patients with human immunodeficiency virus infection. National Institute of Allergy and Infectious Diseases AIDS Clinical Trials Group. N Engl J Med. 1997 May 22;336(21):1487-93. doi: 10.1056/NEJM199705223362103. PMID 9154767
- [Background] Bauditz J, Schachschal G, Wedel S, Lochs H. Thalidomide for treatment of severe intestinal bleeding. Gut. 2004 Apr;53(4):609-12. doi: 10.1136/gut.2003.029710. PMID 15016759
- See also: Approved drug page at FDA's Drugs@FDA web site — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Overview&D...
- See also: Protocol of previous open-label, randomised, iron-controlled study of long-term effects of thalidomide for recurrent gastrointestinal bleeding due to vascular malformation — http://clinicaltrials.gov/ct2/show/NCT00964496?term=thalidomide&rank=2Edit&uid=U0000WPJ&ts=77&cx=-wcbp7